CLINICAL TRIAL: NCT03949543
Title: A Randomised Controlled Trial of Meal Timing as an Acute Modifier of the Gut Microbiota and the Cardiometabolic Health of the Host.
Brief Title: The Timing of Main Meal Consumption Effect on Gut Microbiota and Host
Acronym: TIMC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Dr Konstantinos Gerasimidis, Senior Lecturer in Clinical Nutrition, University of Glasgow
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 200170046
Record Dates: First submitted 2019-05-09; First posted 2019-05-14 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Feeding Behavior; Gastrointestinal Microbiome; Diet; Meal Time
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Adult Participants A (Experimental): Participants who will get two interventional diets, for 7 days each, but allocated to start with large lunch intervention
  Interventions: Other: Large Lunch Intervention; Other: Large Dinner Intervention
- Healthy Adult Participants B (Experimental): Participants who will get two interventional diets, for 7 days each, but allocated to start with large dinner intervention
  Interventions: Other: Large Lunch Intervention; Other: Large Dinner Intervention

INTERVENTIONS:
Other: Large Lunch Intervention — Participants were asked to consume 60% of their daily energy requirements as lunch, between 12:30 and 13:30. Breakfast accounted for 15% of their total daily energy, a morning and evening snack for 5%. 15% was given for light meal either as dinner.
Other: Large Dinner Intervention — Participants were asked to consume 60% of their daily energy requirements as dinner, between 19:30 and 20:30, each day during their two dietary interventions. Breakfast accounted for 15% of their total daily energy, a morning and evening snack for 5%. 15% was given for light meal either as lunch.

SUMMARY:
The interplay between diet and the gut microbiota has been implicated in the onset of cardiovascular disease. The gut microbiota displays diurnal rhythms, which may be influenced by meal timing. This study aimed to investigate the effect of main meal consumption timing on the microbiota and the cardiometabolic factors of the host using a cross-over RCT in healthy adults

The main outcome measurements will be: a) changes in gut microbiota composition based on 16S rRNA gene amplicon sequencing and shotgun metagenomics, b) changes in bacterial functional capacity) and urinary/faecal metabolomics, c) changes in targeted bacterial metabolites, d)Inflammatory markers

The aim of this study is to explore the effect of the timing of main meal consumption on gut microbiota and immune response in healthy adults.

DETAILED DESCRIPTION:
This study will be an open-label, cross-over RCT in healthy adults. Healthy adult (>18 y) participants will be recruited from the community by means of an advertisement leaflet (see associated supporting document-"Advertisement flyer") and word of mouth. The researcher will arrange a meeting with those expressing an interest about the study. The researcher will collect demographic information (e.g. age and gender) and ask the subjects whether they suffer from any acute or chronic illness (defined as illness which requires regular visits to health services) (see associated supporting document-"Health Questionnaire"). If they suffer from a chronic illness they will be excluded. Other exclusion criteria include history of previous of major gut surgery, unstable weight, use of antibiotics or steroids the last 3 months. Participants will be informed about the study at Human Nutrition, New Lister Building, Glasgow Royal Infirmary, or at the University of Glasgow main campus social areas (e.g. Gilchrist). No children will be recruited. Subjects who have expressed an interest about the study but are not suitable to participate will be acknowledged and will receive an explanation as to why they have been excluded.

Following informed written consent, participants will be randomly allocated to intervention groups using the MS Excel "rand()" function. Women will start their intervention on the same phase of their menstrual cycle to avoid the effect of hormonal changes on study outcome.

Dietary interventions: Participants will be asked to undertake two experimental diets. The two dietary interventions are identical with the only difference being the timing of the main meal consumption (dinner and lunch). Participants will follow each diet for a period of one week with a three week washout period between the two interventions. The wash out period aims to drive the gut microbiota characteristics back to baseline levels. The diet will provide the average energy requirements of the participants (Department of Health) and aims to keep participants' weight stable during the study period. All dietary aspects of the study will be designed and supervised by the qualified dietitians/nutritionists, who are members of the research team. Participants will be given a list of meals and snacks to choose from (see associated supporting document-"Food List Preferences"). All meals will be provided to the participants free of charge. Meals will be ordered online by the researchers, using the University of Glasgow Hub, and will be delivered to the participants' residence by the supermarket staff. Weight and height will be measured.

Week 1 Participants will follow a structured diet containing meals of their choice for a week. The participants will select these meals from a list which the researcher will provide to them. The timing of the meal will be specified and the participants will have to complete their meals within 25±5 minutes. The participants will be given written instructions on how to follow the diet (see associated supporting document-"Instruction Sheet" & "Participant Study Calendar"). Participants will provide all faecal samples produced during days from noon of day 5 to noon of day 8. Fasted blood (6 ml) and urine samples will be collected the day after the end of the Week 1 intervention (i.e. day 8). These will be collected at the Human Nutrition laboratory, at the New Lister Building, Glasgow Royal Infirmary. Weight and height measurements will be repeated.

Week 2, 3 & 4 During the wash out period, the participants will follow their habitual diet and no research intervention will take place.

Week 5 This will be replication of the dietary intervention and sample collection at Week 1. The only difference is that lunch meal from Week 1 will swap to dinners in Week 5.

Diet compliance: Over the course of the two experimental diets compliance will be monitored by asking participants to complete a "checklist" with their prescribed diet (see associated supporting document-"Compliance Questionnaire"). A gentle reminder call or text will be sent to the participants every 3 days to increase participants' motivation and compliance on the diets.

Sample collection & analysis: Fresh faecal and urine samples will be collected as described above. The main outcome measurements will be: a) changes in gut microbiota composition based on 16S rRNA gene amplicon sequencing and shotgun metagenomics, b) changes in bacterial functional capacity (whole genome shotgun metagenomics) and urinary/faecal metabolomics, c) changes in targeted bacterial metabolites (short chain fatty acids, sulphide, ammonia, lactate, succinate, ethanol). Blood lipids, appetite hormones, adipokines, and inflammatory markers will be measured using ELISA kits. Stool samples will be collected from participants' homes or delivered to the lab by pre-paid taxi.

Detailed analysis: Genomic DNA will be extracted by the faecal samples using in-house developed assays. The sample will be tested for purity on 1% Agarose gel and the concentration of nucleic acids will be measured with Nanodrop. Amplification of the V4 region of the 16S rRNA gene will be performed in house using PCR and High Fidelity Mastermix and Golay Barcodes. The pooled sample will be sent to the University of Birmingham for 250 bp pair-end sequencing on MiSeq. The data will be analysed by Dr Gerasimidis PDRA in Bioinfomatics. Similarly measurements of SCFA will be performed in acidified ether extracts using Gas Chromatography equipped with an FID detector. Quantification will be performed against authentic standards. Other bacterial metabolites and cardiovascular markers will be assayed with colorometric and enzymatic assays and commercially available ELISA kits as these have been reported previously. https://www.ncbi.nlm.nih.gov/pubmed/28318688 and https://www.ncbi.nlm.nih.gov/pubmed/26119811

Power calculation: An accurate power calculation is impossible to compute due to lack of pilot data. Based on a similar study for a mean difference of 5.4 μmol/g of faecal acetate (SD=5) and 80% power, 20 participants are required. Power calculation will be revised following recruitment and study completion of the first 7 participants.

ELIGIBILITY:
Inclusion Criteria:

1) Healthy adult people

Exclusion Criteria:

1. History of gut surgery
2. Use of antibiotics or steroids the last 3 months
3. Positive or negative energy balance (recent weight gain or loss, ±2 Kg the past month)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2018-05-28 (Actual); Study Completion 2018-05-28 (Actual)

PRIMARY OUTCOMES:
Gut microbiome alpha diversity | 7 days post-intervention
  Shannon diversity index
Faecal short chain fatty acids | 7 days post-intervention
  Short chain fatty acids (umol/g)

SECONDARY OUTCOMES:
HDL | 7 days post-intervention
  mmol/L
LDL | 7 days post-intervention
  mmol/L
Triglycerides | 7 days post-intervention
  mmol/L
Glucose | 7 days post-intervention
  mmol/L
Insulin | 7 days post-intervention
  mU/L
IL-6 | 7 days post-intervention
  pg/mL
tnf alpha | 7 days post-intervention
  pg/mL

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Gerasimidis, BSc MSc PhD, Principal Investigator — University of Glasgow
Locations (1):
- School of Medicine, University of Glasgow / New Lister Building, Glasgow Royal Infirmary, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No